CLINICAL TRIAL: NCT06321484
Title: A Phase 1b Study of Cytokine-Induced Memory Like (CIML) Natural Killer (NK) Cell Therapy in Recurrent Ovarian Cancer
Brief Title: Intraperitoneal Cytokine-Induced Memory Like (CIML) Natural Killer (NK) Cells in Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: ImmunityBio, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Porter, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-493
Record Dates: First submitted 2023-10-30; First posted 2024-03-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Platinum-resistant Ovarian Cancer; Recurrent Ovary Cancer; Ovarian Cancer; Ovarian Carcinoma; Ovarian Carcinoma, Recurrent
Keywords: Platinum-Resistant Ovarian Cancer; Recurrent Ovary Cancer; Ovarian Cancer; Ovarian Carcinoma; Ovarian Carcinoma, Recurrent
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Level 0 (Experimental): Participants will be enrolled in a staggered fashion into a 3+3 dose de-escalation per protocol to establish a maximum tolerated dose (MTD). Dosage will start at dose level 0.
  * Baseline visit.
  * MRIs, PET scans, and/or CT scans every 8 weeks.
  * Cycle 0:
    * Day -7 of 8 day cycle: Apheresis for autologous NK cell collection.
    * Days -6 through -2 of 8 day cycle: Predetermined dose of lymphodepleting chemotherapy per protocol.
    * Days -5 through -4 of 8 day cycle:
      * Predetermined dose of lymphodepleting chemotherapy per protocol.
      * Predetermined dose of premedication per institutional standards.
    * Day 0 of 8 day cycle:
      * Predetermined dose of CIML NK cells once
      * Subcutaneous low-dose IL-2 once
  * Cycle 1:
    - Days 2-8: Subcutaneous low-dose IL-2 every other day for 4 additional doses
  * Off-Treatment:
    * Long-term follow up for 5 years after last CIML NK cell infusion.
  Interventions: Biological: Cytokine-Induced Memory-like Natural Killer Cells; Drug: Interleukin 2
- Dose Level -1 (Experimental): 3+3 de-escalation to dose level -1 per protocol if DLTs occur in Cohort 1 dose Level 0.
  * Baseline visit.
  * MRIs, PET scans, and/or CT scans every 8 weeks.
  * Cycle 0:
    * Day -7 of 8 day cycle: Apheresis for autologous NK cell collection.
    * Days -6 through -2 of 8 day cycle: Predetermined dose of lymphodepleting chemotherapy per protocol.
    * Days -5 through -4 of 8 day cycle:
      * Predetermined dose of lymphodepleting chemotherapy per protocol.
      * Predetermined dose of premedication per institutional standards.
    * Day 0 of 8 day cycle:
      * Predetermined dose of CIML NK cells once
      * Subcutaneous low-dose IL-2 once
  * Cycle 1:
    - Days 2-8: Subcutaneous low-dose IL-2 every other day for 4 additional doses
  * Off-Treatment:
    * Long-term follow up for 5 years after last CIML NK cell infusion.
  Interventions: Biological: Cytokine-Induced Memory-like Natural Killer Cells; Drug: Interleukin 2

INTERVENTIONS:
Biological: Cytokine-Induced Memory-like Natural Killer Cells — Cytokine Induced Memory-like Natural Killer (CIML NK) Cells Autologous, cytokine induced memory-like natural killer cells, via intraperitoneal (IP) infusion per protocol.
  Other Names: CIML NK Cells
Drug: Interleukin 2 — Low dose subcutaneous IL-2 will be administered every other day for 5 doses after CIML NK cell infusion

SUMMARY:
The goal of this research study is to evaluate the safety and effectiveness of the use of cytokine-induced memory-like (CIML) natural killer (NK) cell therapy in recurrent, high grade ovarian cancer (HGOC).

Names of the study therapies involved in this study are:

CIML NK (cellular therapy) Interleukin-2 (IL-2)

DETAILED DESCRIPTION:
This is an open-label, single site, phase 1b study to evaluate the safety and effectiveness of the use of cytokine-induced memory-like (CIML) natural killer (NK) cell therapy in recurrent, high grade ovarian cancer.

Participants will be enrolled to test the safety of intraperitoneal CIML NK cell therapy

The U.S. Food and Drug Administration (FDA) has not approved CIML NK cell therapy as a treatment for recurrent, high grade ovarian cancer.

The research study procedures include screening for eligibility, collection of natural killer (NK) cells in a process called leukapheresis, lymphodepleting chemotherapy, infusion of CIML NK cell therapy into the abdominal cavity (intraperitoneal), administration of low-dose IL-2, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET) scans, blood tests, urine tests, electrocardiograms (ECGs), and echocardiograms.

Participants in this research study will be followed for up to for 5 years after start of study treatment.

It is expected that about 12-18 people will take part in this research study.

The PHASE ONE Foundation Community Research Grant is providing funding for this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed recurrent epithelial ovarian cancer. Eligible histologies include high grade endometrioid or high grade serous ovarian carcinoma.
* Participants must have measurable cancer defined by RECIST 1.1 criteria. Recurrent cancer must be isolated to the abdomen or pelvis with no obvious extra-abdominal metastases via radiographic imaging or physical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Patients must have received at least 1 lines of prior systemic therapy and be deemed platinum resistant/intolerant by their treating oncologist. Patients with germline or somatic BRCA1 or BRCA2 mutations must have received prior PARP inhibitor therapy as maintenance or treatment. Prior receipt of immune checkpoint blockade is allowed if grade 3 or higher toxicities were not experienced.
* Age ≥18 years and <85 years old. Because no dosing or adverse event data are currently available on the use of CIML NK cells in combination with N-803 in participants <18 years of age, children are excluded from this study.
* ECOG performance status of 0 or 1 (see Appendix A).
* Participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥75,000/mcL
  * AST(SGOT)/ALT(SGPT) ≤3 x institutional ULN
  * Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * Serum creatinine ≤ 2.0 mg/dL OR glomerular filtration rate (GFR) ≥40 mL/min/1.73 m2
  * Oxygen saturation: ≥ 90% on room air
  * Left ventricular ejection fraction (cardiac function) ≥ 40%
  * No laboratory evidence of ongoing hemolysis in opinion of investigator
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Physician assessment indicating the patient would be able to tolerate undergoing a brief procedure for placement of an intraperitoneal port for NK cell infusion.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)
* The effects of CIML NK cells and N-803 on the developing human fetus are unknown. For this reason and because CIML NK cells and N-803 are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Participants with distant metastasis outside of the abdominopelvic cavity (e.g., central nervous system, pulmonary, osseous, etc.) whereby intraperitoneal treatment would potentially have minimal effect.
* Participants who have had anti-tumor chemotherapy or other investigational agents within two weeks prior to NK cell infusion (6 weeks for nitrosoureas or mitomycin C), or immunotherapy within 6 weeks prior, or those who have not recovered from adverse events due to agents administered more than two weeks prior. The intent of the language is to ensure that anti-tumor chemotherapy or other investigational agents are not administered to subjects within the specified window since the can potentially affect NK cell activity. Therefore, the washout period is defined by time from NK cell infusion and not patient enrollment. During eligibility confirmation from the study team is requested to confirm that according to the planned NK cell dosing schedule, the washout period should be completed, based on each drug class.
* Participants with a bowel obstruction within the last 3 months or high risk for bowel obstruction (in the opinion of the investigator) or current need for parenteral nutrition or dependence on intravenous fluids.
* Participants who are receiving any other investigational agents.
* Solid organ transplant (allograft) recipients.
* Participants with known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of the first dose of study treatment with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other non-invasive or indolent malignancy, or cancers from which the patient has been disease-free for > 1 year after treatment with curative intent.
* History of severe or anaphylactic allergic reactions attributed to compounds of similar chemical or biologic composition to N-803 or any of the other agents used in study.
* For patients with prior exposure to check point inhibitor therapy, those with a prior history of immune-related toxicity during immune therapy that resulted in permanent discontinuation of therapy (as recommended per product label or consensus guidelines) OR any immune-related toxicity requiring intensive or prolonged immunosuppression to manage (with the exception of endocrinopathy that is well-controlled on replacement hormones) are excluded.
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [Wegener's granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g., GuillainBarre syndrome and myasthenia gravis). Patients with Hashimoto thyroiditis are eligible.
* Systemic corticosteroid therapy (> 10 mg of prednisone or equivalent dose of systemic steroids for at least 4 weeks prior to NK cell infusion). The intent of this language is to ensure that systemic steroids are not administered to subjects within the specified window since this can potentially affect NK cell activity. Therefore, the washout period is defined by time from NK cell infusion and not patient enrollment. During eligibility confirmation the study team is requested to confirm that according to the planned NK cell dosing schedule, the washout period should be completed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the unknown teratogenic risk of CIML NK cells and NIZ985 and with the potential for teratogenic or abortifacient effects by fludarabine/cyclophosphamide chemotherapy regimen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CIML NK cells and NIZ985, breastfeeding should be discontinued if the mother is treated on this study.
* HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions with anti-retroviral agents used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high-risk of lethal treatment-related hepatotoxicity in the setting of marrow suppression. Known non-infectious pneumonitis or any history of interstitial lung disease.
* Receipt of a live vaccine within 30 days of start of study treatment. During eligibility confirmation the study team is requested to confirm that according to the planned NK cell dosing schedule, the washout period should be completed.
* Anaphylactic reactions to murine-based antibody therapy or iron dextran as the CIML NK cell product contains similar reagents at end of manufacturing/infusion.
* Prior history of Grade 2 or higher hemolytic anemia (>/= 2g decrease in hemoglobin plus laboratory evidence of hemolysis) from any cause.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Cohort 1) | 60 days
  The MTD of the use of cytokine induced memory-like natural killer (CIML NK) cell therapy is determined by the number of participants who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for DLT definition.
Dose Limiting Toxicity (DLT) (Cohort 1) | 60 days
  A DLT is defined as an adverse event that is related to CIML NK cell therapy with an attribution of possible, probable, or definite, and meets the criteria defined in protocol section 5.4.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 5 years
  ORR is defined as the proportion of participants who achieved partial response or complete response during study treatment based on RECIST 1.1 and immune-related RECIST criteria.
Median Progression Free Survival (PFS) | Up to 5 years
  PFS is defined as the time from registration to the earlier of progression (PD) or death due to any cause based on Kaplan-Meier methodology. Participants alive without disease progression are censored at date of last disease evaluation.
Clinical Benefit Rate (CBR) | Up to 5 years
  CBR is defined as the proportion of participants who achieved a complete response, partial response, or had stable disease for 6 months or more based on RECIST 1.1 and immune-related RECIST criteria.
Duration of Response (DOR) | Up to 5 years
  DOR is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first data that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
6 months Progression Free Survival (PFS6) | 6 months
  PFS6 is the percent probability estimate at 6 months based on the Kaplan-Meier method. PFS is defined as the time from registration to the earlier of progression (PD) or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Porter, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu